CLINICAL TRIAL: NCT01132833
Title: Chemotherapy and Anti-angiogenic Agents- Induced Thrombosis in Cancer.
Brief Title: Biomarkers Related to Thrombosis in Patients With Newly Diagnosed Multiple Myeloma Receiving Chemotherapy
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC 0802; P30CA016086 (NIH); CDR0000674053 (Other: PDQ number)
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Myeloma; Plasma Cell Neoplasm; Thromboembolism
Keywords: thromboembolism; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Thromboembolism | interventions — Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: enzyme-linked immunosorbent assay — Measurement of markers of coagulation and endothelial activation
Other: laboratory biomarker analysis — The PPP will be used for in vitro assays to measure TF activity, coagulation markers and markers of endothelial cell damage
Other: medical chart review — The patient's clinical course with respect to development of venous thromboembolism and response to treatment will be monitored for a total of 3 months from enrollment.

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients receiving chemotherapy may help doctors learn more about the effects of chemotherapy on cells. It may also help doctors understand how patients respond to treatment.

PURPOSE: This research study is studying biomarkers related to thrombosis in patients with newly diagnosed multiple myeloma receiving chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To measure levels of circulating tissue factor (TF) in patients with newly diagnosed multiple myeloma at several time points before, during, and after the administration of chemotherapy and/or antiangiogenic agents.

Secondary

* To measure the correlation of TF with two markers of coagulation activation (i.e., D-dimer, thrombin-antithrombin [TAT] complexes) and two markers of endothelial activation (i.e., soluble E-selectin, soluble thrombomodulin) in these patients.
* To measure and compare (descriptively) our microparticle-associated TF procoagulant activity assay with two other assays using samples from these patients.

OUTLINE: Patients undergo blood sample collection at baseline and then periodically during treatment. Circulating tissue factor (TF) activity levels and coagulation and endothelial activation (by ELISA) are measured. Medical charts are reviewed for sociodemographic and medical information.

After completion of study, patients are followed up for 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed; relapsed, or refractory multiple myeloma

PATIENT CHARACTERISTICS:

* Central venous access devices allowed
* Recruited by the Division of Hematology/Oncology and the Lineberger Comprehensive Cancer Center at the University of North Carolina
* No history of venous thromboembolism
* No hospitalization for > 2 days within the past month
* Not pregnant
* No patient who refuses or is deemed unsuitable for chemotherapy

PRIOR CONCURRENT THERAPY:

* No surgery within the past month

  * Bone marrow biopsies, central venous line placement and diagnostic biopsies by surgery or fine-needle aspiration allowed
* * No concurrent anticoagulation therapy

  * Concurrent antiplatelet agents, such as aspirin and/or clopidogrel, allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed multiple Multiple Myeloma
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2008-12; Primary Completion 2012-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Levels of circulating tissue factor (TF) | 5 years

SECONDARY OUTCOMES:
Alteration in coagulation parameters | 5 years
Correlation of TF with markers of coagulation activation and endothelial activation | 5 years
Incidence of venous thromboembolism | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Mackman, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: web address for Lineberger Comprehensive Cancer Center, UNC — http://www.unclineberger.org
- See also: web address for the National Cancer Institute (NCI) — http://www.cancer.gov